CLINICAL TRIAL: NCT02483897
Title: Effect of Tetracaine on Pain Management and Corneal Healing in Patients With Acute Corneal Abrasion
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: inabililty to recruit at required rate
Sponsor: Queen's University (Other)
Responsible Party: Principal Investigator, Dr. Robert Brison, Principal Investigator, Queen's University
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 6015429
Record Dates: First submitted 2015-06-18; First posted 2015-06-29 (Estimated); Last update posted 2018-06-04 (Actual); Status verified 2018-06

CONDITIONS: Corneal Abrasion
MeSH Terms: conditions — Corneal Injuries | interventions — Tetracaine; Ophthalmic Solutions

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tetracaine 0.5% ophthalmic drops (Experimental): 0.8 mls. drops provided to be used hourly p.r.n. for pain control
  Interventions: Drug: Tetracaine 0.5% ophthalmic drops
- placebo (Normal Saline placebo drops) (Placebo Comparator): 0.8 mls. drops provided to be used hourly p.r.n. for pain control
  Interventions: Drug: Normal Saline placebo drops

INTERVENTIONS:
Drug: Tetracaine 0.5% ophthalmic drops — 0.8 mls. drops provided to be used hourly p.r.n. for pain control
  Arms: Tetracaine 0.5% ophthalmic drops
Drug: Normal Saline placebo drops — 0.8 mls. drops provided to be used hourly p.r.n. for pain control
  Arms: placebo (Normal Saline placebo drops)

SUMMARY:
Corneal abrasions are associated with significant discomfort during a 24-48 hrs healing phase. Current practice guidelines discourage the use of topical anesthetics in treating these patients due to concerns that these medications may prevent proper corneal epithelial healing. These concerns are based primarily on decades old animal based research. However, recent evidence suggests topical anaesthetics are a safe and effective way of managing patient pain in the short term. This study will investigate the effect of topical 0.5% tetracaine on corneal healing and pain management in patients with corneal abrasions in the first 48 hours.

This will be a prospective, double blind, randomized, controlled study of 260 adults with uncomplicated acute corneal injuries presenting to the tertiary acute care settings in Kingston. Patients will be randomly assigned to receive either 0.5% tetracaine or saline in addition to usual care as outpatients. They will be followed through the ophthalmology emergency eye clinic to assess healing at 36-48hrs. after the acute care visit. The primary outcome will be an assessment of pain as measured every 4 hours for 48 hrs. using a 10mm Visual Analogue Scale (VAS). Secondary outcomes will include assessments of corneal healing, use of adjunct pain medications, time lost from work/usual activities, quality of sleep, ability to read and the SF12 quality of life questionnaire.

This study will better inform the safety and effectiveness of short-term tetracaine usage in patients with simple corneal abrasions for optimal treatment of patients in the future.

DETAILED DESCRIPTION:
Corneal abrasions are commonly encountered eye injuries presenting to acute care settings and account for over 10% of new ophthalmological presentations at eye accident departments, primary care offices, and emergency departments. Patients complain of severe eye pain, foreign body sensation, pain with blinking, and photophobia. Corneal abrasions are defects in the epithelial layer that occur secondary to mechanical ocular surface trauma. Common causes of corneal abrasions include fingernail injuries, tree branches, and projectile pieces of metal, wood, or glass that injure or become embedded in the cornea. . Though associated with significant discomfort, the prognosis for simple corneal abrasions is usually excellent, with full recovery within 24-48 hours. Untreated abrasions, particularly those associated with a retained foreign body, can lead to complications such as corneal ulcers, prolonged pain, and visual acuity loss.

Currently, the standard approach to treating corneal abrasions includes removal of the foreign body if present, oral analgesics for pain control, and topical antibiotics. Traditional guidelines by ophthalmologists have advocated against the use of topical anesthetics due to concerns with corneal epithelial healing the potential for patients to miss important clinical clues that indicate the rare development of secondary corneal infection, as well as the potential for longer term misuse leading to severe corneal ulceration and perforation. Previous studies, primarily using animal models, have found a delay in corneal epithelial healing with topical anaesthetics, particularly with repeated and prolonged usage. Several case studies have described impaired corneal epithelial healing and ulceration with the prolonged use and abuse of topical anesthetic drops (0.05% proparacaine HCl). There have been reports of topical anesthetic (TA) induced corneal damage including punctate epitheliopathy, corneal lysis, perforation, persistent epithelial defects, and ocular inflammation. It is thought that local anesthetics inhibit mitosis and cellular migration, preventing proper re-epithelialization of the cornea.

However, in recent years a number of randomized clinical trials and case studies of human subjects have shown that with appropriate application and restricted short term usage, topical anesthetics did not delay wound healing or increase risks of corneal ulceration.

A recent prospective, randomized, double-blind trial looked at the effect of topical anesthetics on epithelial healing and pain management for patients with uncomplicated corneal abrasion. The study included 116 patients presenting to the emergency department who were given either 1% tetracaine HCl or control artificial tears. The study found no change in corneal healing rate or persistent symptoms but little benefit in pain relief as measured at 48 hrs. A previous prospective randomized study comparing 0.05% proparacaine and placebo has shown a significant decrease in reported pain with topical anesthetic use compared to control with no change in corneal healing. Another study evaluating the effect of 1% tetracaine for pain management after photorefractive keratectomy also reported significant pain reduction with topical anesthetic use with no delays in epithelial healing.

Controversy continues to exist over the utility of topical anesthetics in managing pain and their safety in affecting corneal healing. Contemporary studies of short term topical anesthetic use, noted above, have not shown adverse effects on healing. Differential effects on pain management have been found. Yet the investigators believe the Waldman study measured pain at a delayed time when the abrasion would be expected to have healed. Clinicians in Queen's Department of Emergency Medicine do not generally prescribe topical anesthetics for corneal abrasions and believe that evidence demonstrating their efficacy and safety would change practice patterns for the benefit of patients with these injuries and those in other centres. The investigators also hope that this study will better address problems of inadequate participant enrollment and retention that previous studies have encountered.

1.3 - Research Question In adult emergency department patients with acute corneal abrasions, is the application of 0.5% tetracaine effective in the short-term management of pain while not being associated with adverse effects on healing?

1.4 - Hypothesis Based on the review of existing literature on the effects of topical anesthetics, the investigators hypothesize that short-term and controlled usage of tetracaine will be an effective way in managing patient pain and will not affect corneal healing.

ELIGIBILITY:
Inclusion Criteria:

* Patients (>18yo) coming in with acute (<24 hours) simple uncomplicated corneal abrasions.

Exclusion Criteria:

1. Patients with frankly contaminated wound, corneal foreign body, or epithelial defect secondary to contact lens wear
2. History of comorbid eye conditions including eye surgery within the past month and glaucoma.
3. Involvement of both eyes
4. Allergy to tetracaine or any of the substances used in the study
5. Unable to provide consent.
6. Unable to come for follow-up.
7. Patients with a past history of corneal injury infection or surgery will undergo a screening test of the corneal sensation. If a diminished or absent sensation is found, the patient will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-06; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
pain control as measured by visual analogue score | at 12 hours post baseline
  10 cm. VAS scale

SECONDARY OUTCOMES:
Compound Outcome comprised of Number of Participants with one or more of listed adverse outcomes including: anaphylactic reaction, infectious infiltrate, stromal/ring infiltrate, corneal ulceration, hypopyon, abrasion size not decreasing | at 36-48 hour follow up appointment
  adverse outcome measure

REFERENCES:
- [Derived] Algarni AM, Guyatt GH, Turner A, Alamri S. Antibiotic prophylaxis for corneal abrasion. Cochrane Database Syst Rev. 2022 May 27;5(5):CD014617. doi: 10.1002/14651858.CD014617.pub2. PMID 35622535